CLINICAL TRIAL: NCT00878748
Title: An Open Label, Prospective and Multi-center Recurrence Prevention Study With Effexor XR in MDD Patients in China
Brief Title: Study Evaluating Effexor XR in Chinese Subjects With Major Depressive Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0600X1-4434
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Effexor XR
  Interventions: Drug: Effexor XR
- B (Other): Effexor XR discontinue
  Interventions: Other: Effexor XR discontinue

INTERVENTIONS:
Drug: Effexor XR
  Arms: A
Other: Effexor XR discontinue
  Arms: B

SUMMARY:
This primary purpose of this study is to assess the efficacy and safety of Effexor XR in preventing recurrence in Chinese patients with recurrent major depressive disorder (MDD) following a 1-year maintenance treatment after an 8-week acute treatment and a 6-month continuation treatment phases. The study will also collect data on the prevalence and pattern of co-morbid anxiety and somatic symptoms and their impact on the recurrence of depression.

ELIGIBILITY:
Inclusion criteria: 1. Males or females, 18 years of age or more; 2. Outpatients; 3. Major depressive disorder based on DSM-IV criteria, with/without current co-morbid anxiety disorder; 4. Has two or more episodes of depression (including the current episode) in the past 5 years, with an interval of at lease 2 months between the end of the previous episode and the beginning of the current episode. 5. The baseline score of 17-item Hamilton Rating Scale for Depression (HAM-D)>=17; 6 If female of childbearing potential, have a negative urine pregnancy test at baseline, if appropriate, and use a medically acceptable method of contraception throughout the study.

Exclusion criteria:1.Hypersensitivity to venlafaxine;2.Received venlafaxine treatment before;3.Clinically significant renal or hepatic disease or any other medical disease that, in the opinion of the investigator, might compromise the study, including seizure disorder (with the exception of a single childhood febrile seizure); 4.Alcohol or drug abuse within the last year;5.A recent history of myocardial infarction or unstable heart disease (within 6 months of baseline);6.Bipolar disorder;7.For female, known or suspected pregnancy or breast feeding;8.Use of a monoamine oxidize inhibitor (MAOI) within 14 days of baseline; use of any investigational drug within 30 days of baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
time from entering maintenance phase to recurrence of major depression | 12 months

SECONDARY OUTCOMES:
Patient Health Questionnaire(PHQ-15),Clinical Global Impressions(CGI),Visual Analogue Scale(VAS),Short Form Health Survey(SF-36) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer